CLINICAL TRIAL: NCT01910909
Title: Effectiveness and Safety of the Stereotactic Body Radiation Therapy for Hepatocellular Carcinoma: Prospective Phase II Trial
Brief Title: Stereotactic Body Radiotherapy for Unresectable Hepatocellular Carcinoma
Acronym: SBRT for HCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Park Hee Chul, Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-06-005-001
Record Dates: First submitted 2013-07-17; First posted 2013-07-30 (Estimated); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Localized Non-Resectable Adult Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; unresectable; small size; Stereotactic body radiotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiosurgery

ARMS (1):
- Stereotactic body radiotherapy (Experimental): Stereotactic body radiotherapy 60 Gy/3 fraction standard dose The highest allowable dose with maintain normal tissue constraints
  Interventions: Radiation: Stereotactic body radiotherapy

INTERVENTIONS:
Radiation: Stereotactic body radiotherapy — Respiration training will be done on the day that patient decided participate this study with wearing video goggle and headphone assisted respiration by visual and voice. Four dimensional CT simulation with wearing video goggle and headphone assisted respiration by visual and voice and real time position management system (PRM) signal will be adopted. Planning MRI with diffusion image also be acquired in same condition with CT simulation. SBRT will be delivered daily 20 Gy for 3 fractions.

SUMMARY:
1. Background 1.1. Hepatocellular carcinoma (HCC) HCC is the third most common cause of cancer death globally. It is also the second cause of cancer mortality in Korea, despite the incidence of HCC was fifth. The most important cause of this discrepancy is connected with the fact that the significant portion of the HCC is detected as unresectable status.

1.2. Standard treatment of the HCC At the point of HCC diagnosis, only 30% of the patients could receive standard curative treatment, like resection, liver transplantation, and radiofrequency ablation (RFA). Transcatheter arterial chemoembolization (TACE) has been shown in randomized trials to improve survival compared with symptomatic therapy alone, in the patients without macrovascular involvement, extrahepatic disease and tumor related symptoms. However, in the recent review of TACE, TACE might be contraindicate or not recommended in the patients who showed vascular tumor invasion, more than 10 cm size, poor portal blood flow and/or repeated poor response.

Recently, Sorafenib, which is one of the target agents, showed survival advantage on unresectable HCC patients in two randomized study. In those study, sorafenib improved approximately three month overall survival increment, however, the median survival duration was only 10.7 months in experiment group (received sorafenib), and even 6.5 months in Asian-Pacific trial. Additionally, the possibility that sorafenib effect could be reduced in the patients had hepatitis B virus (HBV) was suggested in the subgroup analysis.

1.3 Radiation therapy (RT) for the HCC The use of RT in HCC is increased with the radiation technological advances. In the unresectable patients, RT showed 50 to 60% response rate with the dose response relationship. Recently, stereotactic body radiation therapy (SBRT) showed excellent local control and comparable survival rate in thoracic tumor. In the HCC, SBRT also showed 75 to 100% local control rate without significant elevation of the toxicities. One study reported that 24 to 54 Gy SBRT achieved 87% 1year local control and 17 months overall survival. The standard treatment of unresectable HCC is sorafenib, but Korean Liver Cancer Study Group (KLCSG) recommend RT as an option in localized unresectable HCC. Furthermore, Radiation Therapy Oncology Group (RTOG) started randomized trial to confirm the effect of SBRT in unresectable HCC (RTOG 1112).

Investigators previously reported the retrospective result that the higher dose SBRT achieved 2 year overall survival 87.9% and local control 85% in the patient who showed less than 5 cm solitary HCC without portal vein involvement.

Based on those studies, we start this prospective study to evaluate the effectiveness and adverse event of SBRT in the patients who had solitary 3 cm or less size HCC without extrahepatic lesion and vascular involvement.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a diagnosis of HCC by at least one criterion listed below (KLCSG guideline 2009) 1.1 Pathologically (histologically or cytologically) proven diagnosis of HCC 1.2 Liver nodule in high risk group 1.2.1 If alpha feto protein (AFP)≥200 ng/mL , ≥ 1 typical HCC enhancing pattern on dynamic contrast enhanced CT or MRI 1.2.2 If AFP<200 ng/mL, ≥2 typical HCC enhancing pattern on dynamic contrast enhanced CT, MRI, and angiography 1.3 ≥ 2 cm nodule in liver cirrhosis (LC), ≥ 1 typical HCC enhancing pattern on dynamic contrast enhanced CT or MRI
2. Eastern cooperative oncology group performance status 0 or 1
3. Size of the HCC ≤ 3 cm or less
4. Age ≥ 20
5. Unsuitable for resection or transplant or RFA
6. Unsuitable for or refractory to TACE or drug eluting beads (DEB)
7. Agreement of study-specific informed consent
8. Assessment by radiation oncologist and medical oncologist or hepatologist within 28 days prior to study entry?
9. Child-Pugh score A within 14 days prior to study entry
10. normal liver (Liver minus gross tumor volume) ≥ 700 cc
11. Target is only one viable hepatocellular carcinoma
12. Blood work requirements

    * Absolute neutrophil count (ANC) ≥ 1,500 /mm3, Platelet ≥ 70,000/mm3, Hgb ≥ 8 g/dl
    * Liver function test (LFT): T. bilirubin<3.0 mg/dL, International normalized ratio (INR) < 1.7, Albumin ≥ 2.8g/dL, Aspartate aminotransferase (AST)/Alanine aminotransferase (ALT)< 6 X normal
    * Serum creatinine < 1.5 X normal, or Creatinine clearance rate ≥ 60 mL/min
13. Male, consent contraception at least 6 months Childbearing potential woman, consent contraception at least 6 months
14. Life expectancy more than 12 weeks
15. Stable breathing more than 10 minutes
16. Consent to fiducial marker insertion ( if needed )

Exclusion Criteria:

1. Extrahepatic metastasis or malignant nodes
2. Pregnant and/or breastfeeding woman
3. Macroscopic vascular tumor involvement
4. Previous upper abdominal RT history
5. Uncontrolled active co-morbidity

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the SBRT effect on local progression free survival rate | Radiologic response will be evaluated at 3 month.
  Radiologic response will be evaluated at 1, 3 month after SBRT, and then every 3 month imaging follow up will be continued. Local progression will be defined by modified Modified response evaluation criteria for solid tumor (mRECIST). Local progression was defined as 20% or more size increase of contrast enhanced primary lesion or new contrast enhanced lesion in planning target volume.
To evaluate the SBRT effect on adverse events | Adverse events will be evaluated at 3 month after SBRT.
  Adverse events will be evaluated at 1 and 3 month after SBRT, and then every 3 month follow up will be continued.. Adverse event will be evaluated with common terminology criteria for adverse events (CTCAE version 4.0) during follow up.

SECONDARY OUTCOMES:
To determine the SBRT objective response rate | Response will be evaluated at 3 month
To measure the time to local tumor progression | Response will be evaluated at 3 month after SBRT.
  Response will be evaluated at 3 month after SBRT, then every 3 month follow up with imaging will be continued. mRECIST will be used to define local tumor progression.
To measure the overall survival | Survival will be evaluated at 3 month after SBRT.
  Survival will be evaluated at 3 month after SBRT, then every 3 month follow up will be continued. Overall survival will be measured from the data of SBRT start to the date of death or to the date of last follow up visit.
To measure the progression free survival | Response will be evaluated at 3 month after SBRT.
  Response will be evaluated at 3 month after SBRT, then every 3 month follow up with imaging will be continued. mRECIST will be used to define response. Progression free survival will be measured from the date of SBRT to the date of progression recognition or to the date of lat follow up visit.

OTHER OUTCOMES:
Quality of life(QOL)change before and after RT | QoL will be assessed before, and 1, 3, 6 months after SBRT.
  To measure the quality of life(QOL) before and after RT, European Organization for Research and Treatment of Cancer (EORTC) core Quality of Life Questionnaire (QLQ)-C30, Functional Assessment of Cancer Therapy-Hepatobiliary (FACT-Hep) will be used. Before simulation of RT, baseline QOL assessment will be obtained, then QOL will be assessed at 1, 3, 6 months after RT, before physician interview.
RT response prediction probability evaluation by diffusion-weighted (DW) MRI and positron emission tomography | At 1 month after RT

CONTACTS AND LOCATIONS:
Overall Officials: Hee Chul Park, M.D., Ph.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea